CLINICAL TRIAL: NCT05094310
Title: Genetic Predictors of Response to Acupuncture for Cancer-related Fatigue Among Breast Cancer Patients After Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHQU-2021007
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
Keywords: Single nucleotide polymorphisms; Breast Cancer; Cancer-related fatigue; Acupuncture
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture group (Experimental): Patients with breast cancer who experienced fatigue were measured by the Brief Fatigue Inventory(BFI) scale and other Fatigue related questionnaire. Breast cancer patients diagnosed with cancer related fatigue are included in our clinical study，and those patients will receive acupuncture treatment. The position of acupuncture refers to the principle of acupuncture treatment of traditional Chinese medicine. According to ICD-10-CD code R53.0, the diagnosis of CRF is determined by the experience of diminished energy or other physical and psychological symptoms every day or almost every day for two consecutive weeks in the past month. We collected patients' blood to detect fatigue related SNP.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Patients with breast cancer who experienced fatigue were measured by the Brief Fatigue Inventory(BFI) scale and other Fatigue related questionnaire. Breast cancer patients diagnosed with cancer related fatigue are included in our clinical study，and those patients will receive acupuncture treatment. The position of acupuncture refers to the principle of acupuncture treatment of traditional Chinese medicine. According to ICD-10-CD code R53.0, the diagnosis of CRF is determined by the experience of diminished energy or other physical and psychological symptoms every day or almost every day for two consecutive weeks in the past month. We collected patients' blood to detect fatigue related SNP.

SUMMARY:
Genetic predictors of response to acupuncture for cancer-related fatigue among breast cancer patients after chemotherapy.

DETAILED DESCRIPTION:
Cancer related fatigue(CRF) in patients with breast cancer has a great impact on their quality of life and treatment compliance. Many studies suggest that acupuncture has certain therapeutic effects on fatigue. In this clinical trial, we treated patients with acupuncture to alleviate their fatigue symptoms. Currently, studies have shown that cancer related fatigue in breast cancer patients is related to some biological factors. While acupuncture is used to treat fatigue, we will collect blood samples from patients for fatigue related single nucleotide polymorphisms（SNP）.

Based on CRF related biological factors, our study aims to screen SNPs that related to CRF related biological factors to guide electroacupuncture in the treatment of cancer-related fatigue and establish a prognostic model.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was diagnosed with breast cancer.;
2. Breast cancer patients diagnosed with cancer related fatigue are included in our clinical study;
3. Voluntarily participate in the clinical trial and sign the informed consent form after informed consent (patients voluntarily accept the treatment and give informed consent);
4. Patients with previous local recurrence were eligible, but not patients with distant metastasis；
5. The basic indexes were consistent, and the blood routine and ECG were normal.

Exclusion Criteria:

1. The exclusion criteria were patients with needle phobia;
2. Low platelet count (<50 000); co-morbidity with a bleeding disorder; co-morbidity with thyroid dysfunction; pregnancy; haemoglobin levels <10 g/dl and haematocrit <30; anaemia on active pharmacological treatment or receiving blood transfusion or steroids；
3. Life expectancy <6 months；
4. lymphoedematous limbs.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Difference of BFI score change after treatment | 2 years
  Brief Fatigue Inventory（ BFI）is a nine item scale used to evaluate the intensity of fatigue and the interference of fatigue to normal activities. The classification of fatigue severity is: Mild fatigue (1-3), Moderate fatigue (4-6) and Severe fatigue (7-10).

SECONDARY OUTCOMES:
Side effects related to electroacupuncture | 2 years
  Side effects related to electroacupuncture

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: No